CLINICAL TRIAL: NCT00564772
Title: An Open-Label, Sequential, 3-Period Study to Evaluate Pharmacokinetics of Coadministered Raltegravir (Isentress) and Lopinavir-Ritonavir (Kaletra) in Healthy Adults
Brief Title: Raltegravir Kaletra Pharmacokinetics
Acronym: RAL-KAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 78958; Allina IRB No. 2366-1; Prism Research No. 714; FDA IND No. 78958
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: raltegravir; lopinavir; ritonavir; pharmacokinetics
MeSH Terms: interventions — Raltegravir Potassium; Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Experimental): all subjects dosed the same
  Interventions: Drug: Raltegravir, lopinavir, ritonavir

INTERVENTIONS:
Drug: Raltegravir, lopinavir, ritonavir — 4 days of raltegravir, then 10 days of Kaletra, then 4 days of both with 12 PK sampling at the end of each period.
  Other Names: Isentress; Kaletra

SUMMARY:
This will be an open-label, 3-period, fixed sequence study in young, healthy, male and female subjects of the pharmacokinetic interaction between raltegravir and Kaletra.

DETAILED DESCRIPTION:
This will be an open-label, 3-period, fixed sequence study in young, healthy, male and female subjects. The initial cohort, to be studied simultaneously, will be 15 subjects with intention to collect complete data from 12 subjects. Replacements will be subsequently enrolled if necessary. Subjects will be reimbursed.

The periods will be

* Period 1: Raltegravir (RAL) 400 mg q12h for 4 days (7 doses of RAL).
* Period 2: Kaletra 200 mg 2 pills bid for 10 days (19 doses of Kaletra).
* Period 3: both regimens for 4 days (7 doses of both drugs). All morning doses will be observed at Prism Research, Inc. Evening doses will be distributed each morning. 12 hour PK studies will be done on the last day of each period. Specimens will be obtained 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours after the morning dose of the last dosing day of each period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male or female, age 18-55.
* Anti-HIV, anti-HCV, HBsAg negative.
* Normal history and physical at screening.
* Normal complete blood count, creatinine and ALT at screening.
* Negative urine pregnancy test at screening.
* BMI 18-30.

Exclusion Criteria:

* Donated blood in the month before Day 1.
* Participated in another research study in the month before Day 1.
* Tobacco use in the 3 months before Day 1, unwillingness to avoid tobacco use during the study.
* Use of any illegal drug in the year before Day 1, positive drug screen for an illegal drug at screening.
* Unwillingness to restrict coffee use to 6 or fewer cups of coffee during the study.
* Unwillingness on the part of fertile female subjects to be abstinent or to use two effective birth control methods, one of which is a barrier method, for any vaginal intercourse.
* Unwillingness to avoid use of any prescribed medication during the study
* Allergy to RAL, lopinavir or ritonavir.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
drug levels of lopinavir, ritonavir, raltegravir | 2 months

SECONDARY OUTCOMES:
safety | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank S Rhame, MD, Principal Investigator — Allina Hospitals & Clinics
Locations (1):
- Prism Research Inc, Saint Paul, Minnesota, United States